CLINICAL TRIAL: NCT03867045
Title: Development of a Cabozantinib (Cabometyx) Symptom Management Application for Use in Patients With Renal Cancer
Acronym: Cabo App
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study deemed non-essential under COVID pandemic,
Sponsor: Duke University (Other)
Collaborators: Exelixis (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: Pro00086667
Record Dates: First submitted 2019-02-15; First posted 2019-03-07 (Actual); Last update posted 2021-06-14 (Actual); Status verified 2020-11

CONDITIONS: Metastatic Renal Cell Carcinoma Treated With Cabozantinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- mRCC treated with cabozantinib (Experimental): Nine patients with mRCC initiating cabozantinib therapy who meet subject eligibility criteria.
  Interventions: Device: Usability of an electronic symptom management application

INTERVENTIONS:
Device: Usability of an electronic symptom management application — Usability of an electronic symptom management application in a pilot group of patients receiving cabozantinib for mRCC through data analytics and feedback from users

SUMMARY:
The purpose of this study is to develop an on-line electronic symptom management application that can ultimately be used to improve clinical outcomes in patients with mRCC treated with cabozantinib.

DETAILED DESCRIPTION:
This is a single-site, prospective technology-based, clinical trial. Nine patients with mRCC initiating cabozantinib therapy who meet subject eligibility criteria will be enrolled in this study. Subjects will be given an iPOD touch with the symptom monitoring application installed, physical activity and blood pressure monitors. Each patient will be kept on study for the first 12 weeks of therapy with cabozantinib. Subjects on treatment for less than 12 weeks will not be replaced.The symptoms and other data (physical activity, blood pressure) recorded electronically by the patient will be compared to symptoms recorded in the medical record at interval clinic visits.

ELIGIBILITY:
Inclusion Criteria:

Patients > 18 years of age Patients planning to start treatment with cabozantinib therapy for renal cancer.

Technology requirement: The patient will need to have home wireless internet access for use of the software and technology in this study. The patient will need to already have or be willing to set up a Duke MyChart account.

Exclusion Criteria:

Non-English Speaking. Any patient who is not able to comprehend and operate the technology at the discretion of the enrolling provider.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2019-08-21 (Actual); Primary Completion 2019-12-16 (Actual); Study Completion 2019-12-16 (Actual)

PRIMARY OUTCOMES:
Number of comments from participants indicating ease of use of the application. | 12 weeks
  Number of comments from participants indicating ease of use of the application.

SECONDARY OUTCOMES:
Blood pressure (BP) readings measured daily by the BP monitoring device compared with those BP readings measured at interval clinic visits within the first 12 weeks to determine similar detection of symptoms. | 12 weeks
  Blood pressure (BP) readings measured daily by the BP monitoring device compared with those BP readings measured at interval clinic visits within the first 12 weeks to determine similar detection of symptoms.
Movement recorded daily by the activity tracking device compared with ECOG assessment outcomes measured during interval clinic visits within the first 12 weeks to determine similar estimates of activity. | 12 weeks
  Movement recorded daily by the activity tracking device compared with ECOG assessment outcomes measured during interval clinic visits within the first 12 weeks to determine similar estimates of activity.
Number and frequency of adverse symptoms reported in the symptom management application compared with clinical assessment of adverse events recorded at interval clinic visits within the first 12 weeks to determine similar report of adverse symptoms. | 12 weeks
  Number and frequency of adverse symptoms reported in the symptom management application compared with clinical assessment of adverse events recorded at interval clinic visits within the first 12 weeks to determine similar report of adverse symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Sundhar Ramalingam, MD, Principal Investigator — Duke University
Locations (2):
- United States (2):
  - Duke University Medical Center, Durham, North Carolina
  - Duke Raleigh Hospital, Raleigh, North Carolina